CLINICAL TRIAL: NCT02348801
Title: Lifestyle Intervention Strategy to Treat Diabetes in Older Adults
Brief Title: Lifestyle Intervention for Senior Diabetics
Acronym: LISD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: American Diabetes Association (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Principal Investigator, Dennis T. Villareal, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-34800
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; Aging; Overweight
MeSH Terms: conditions — Diabetes Mellitus; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Lifestyle Group (Active Comparator): Group diabetes educations sessions that focus on diet, exercise, and social support.
  Interventions: Behavioral: Healthy lifestyle
- Weight Loss plus Exercise Group (Experimental): Behavioral therapy for weight loss and exercise training
  Interventions: Behavioral: Weight loss and Exercise

INTERVENTIONS:
Behavioral: Weight loss and Exercise — Group behavior therapy sessions designed to acquire positive weight-control skills and attitudes, and practice weight-maintenance skills. A balanced diet will be prescribed to provide a deficit of 500-750 kcal/day from daily energy requirement.
  Exercise sessions of ~90 min duration 15 min warm-up of flexibility exercise, followed by ~30 min of aerobic exercise, and, after a brief rest period, ~30 min of resistance training, and finally ~15 min balance exercise) conducted three times weekly supervised at our exercise facility for first six months, and regular exercises continued at community-fitness centers and at home for the following six months.
  Arms: Weight Loss plus Exercise Group
Behavioral: Healthy lifestyle — Diabetes support and education
  Arms: Healthy Lifestyle Group

SUMMARY:
Older people with diabetes will be assigned to the 1-year lifestyle program or no lifestyle program while continuing usual treatment for diabetes. The lifestyle program will consist of teaching how to practice healthy diet and regular exercise at our facility and continued into the community and home. It is hoped that the results would provide convincing proof about the usefulness of lifestyle change in older patients with diabetes.

DETAILED DESCRIPTION:
Background: Hypothesis: Lifestyle intervention will be highly successful in the population of older adults with diabetes, with resultant significant improvement in glycemic metabolic control mediated by improved insulin action/secretion, accompanied by significant improvements in physical function, cognitive function, and quality-of-life (QOL).

Rationale: Countering the prevailing notion that it is difficult to change lifelong habits, the PI has ample preliminary data showing successful lifestyle change in older adults. A similar lifestyle intervention augmented by motivational interviewing might also be successful in older adults with diabetes with eventual translation to the community- and home-settings.

Aims: In older adults with diabetes and comorbidities, the aims are to: determine the effect of lifestyle intervention on glycemic metabolic control, determine the mechanisms underlying lifestyle-induced changes in glucose homeostasis, and determine the effect of lifestyle intervention on age-relevant health outcomes: physical function, cognitive function, QOL.

Design: Older adults with diabetes and comorbidities will be randomized to center-based lifestyle intervention continued into the community and home vs. healthy-lifestyle control for 1 year.

Relevance to diabetes prevention and treatment: Data from a randomized-controlled trial will provide high-level evidence to convince practitioners to implement lifestyle intervention as the primary therapy for diabetes in older patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be older (age 65-85 years) adults with type 2 diabetes. Diabetes will be determined by self-report with verification (medical records, current treatment, confirmation from health care provider, fasting glucose ≥126 mg/dL, symptoms of hyperglycemia with plasma glucose ≥200 mg/dL or 2-hour plasma glucose ≥200 mg/dL after a 75-g glucose load on at least two occasions, or HbA1C of ≥ 6.5%. All subjects will have a BMI of ≥ 27 kg/m2 and have stable weight (±2 kg) and on stable medications during the last 6 mos.

Exclusion Criteria:

* Volunteers will be excluded if they fail to provide informed consent, have any major comorbid disease that is uncontrolled, or any condition that is likely to limit life span and/or affect the safety of the interventions, or interfere with the conduct of the trial. Examples include: 1) unstable cardiopulmonary disease (e.g. recent MI, unstable angina, stroke within past 3 months) or unstable disease (e.g. Class IV congestive heart failure: 2) severe orthopedic (e.g. awaiting joint replacement) and/or neuromuscular (e.g. multiple sclerosis, amyotrophic lateral sclerosis, active rheumatoid arthritis), 3) significant cognitive impairment, defined as a known diagnosis of dementia or positive screening test for dementia using the Mini-Mental State exam (i.e. MMSE score <24),43 4) cancer requiring treatment in the past 5 years, 5) documented history of pulmonary embolism in the past 6 months, 6) positive exercise stress test for cardiac ischemia, and 7) HbA1c >11%.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | baseline and 12 months

SECONDARY OUTCOMES:
Change in insulin sensitivity | baseline and 12 months
Change in insulin secretion | baseline and 12 months
Change in fasting glucose | baseline and 12 months
Change in adipocytokines and hormones | baseline and 12 months
Change in peak aerobic power | baseline and 12 months
Change in cardiometabolic risk profile | baseline and 12 months
Change in the modified physical performance test | baseline and 12 months
Change in composite cognitive z-score | baseline and 12 months
Change in quality of life | baseline and 12 months
Change in health care utilization | baseline and 12 months
Change in the modified mini-mental state exam | baseline and six months
Change in muscle strength and quality | baseline and 12 months
Change in gait speed | baseline and 12 months
Change in stroop color naming | baseline and 12 months
Change in word list fluency | baseline and 12 months
Change in ray auditory verbal learning test | baseline and 12 months
Change in Trail A./B | baseline and 12 months
Change in Lean body mass | baseline and 12 months
Change in fat mass and visceral fat | baseline and 12 months
Change in bone mineral density | baseline and 12 months
Change in bone metabolism | baseline and 12 months
Change in bone quality | baseline and 12 months
Change in composite cognitive score | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Celli A, Barnouin Y, Jiang B, Blevins D, Colleluori G, Mediwala S, Armamento-Villareal R, Qualls C, Villareal DT. Lifestyle Intervention Strategy to Treat Diabetes in Older Adults: A Randomized Controlled Trial. Diabetes Care. 2022 Sep 1;45(9):1943-1952. doi: 10.2337/dc22-0338. PMID 35880801